CLINICAL TRIAL: NCT06935604
Title: Healing Hearts of Hospitalized Patients: A Randomized, Non-inferiority Study of Virtual Reality Facilitation
Brief Title: Healing Hearts of Hospitalized Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 80473
Record Dates: First submitted 2025-04-12; First posted 2025-04-20 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Pain; Anxiety; Stress; Loneliness
Keywords: Virtual Reality
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR a trained facilitator. (Active Comparator)
  Interventions: Behavioral: VR with a trained facilitator
- VR without a trained facilitator. (Experimental)
  Interventions: Behavioral: VR without a trained facilitator.

INTERVENTIONS:
Behavioral: VR with a trained facilitator — Intervention Group 1 - VR with a facilitator:
  Each participant in the intervention group will undergo a structured VR session, consisting of:
  Duration: 20 minutes Content: Immersive VR experience designed to promote relaxation and reduce pain.
  Facilitator training: The facilitator group will include trained healthcare professionals skilled in VR technology, C-I-CARE, and empathetic patient engagement. All facilitators also complete the Creative & Healing Arts Heart-to-Heart training which includes observation, empathy training, and reflection to support complex communication, and companionship needs of adult patients .
  Arms: VR a trained facilitator.
Behavioral: VR without a trained facilitator. — Intervention Group 2 - VR without an inperson facilitator:
  Each participant in the intervention groups will undergo a structured VR session, consisting of:
  Duration: 20 minutes Content: Immersive VR experience designed to promote relaxation and reduce pain.
  Instructional video: A research assistant will use C-I-CARE to give the patient an instructional video and the headset to engage in the VR technology.
  Patients will take a surveys before and after the intervention
  Arms: VR without a trained facilitator.

SUMMARY:
The study aims to study virtual reality (VR) facilitation with adult inpatients using VR as a way to alter pain perception and reduce emotional distress during their hospitalization. Specifically, this study will evaluate the outcomes of patients who experience VR with and without a trained facilitator as a form of escapism.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and above
* Able to provide informed consent
* Able to follow commands
* Adequate motor skills for upper extremities to operate VR equipment
* Clinically stable
* English speaking
* Willing to engage in VR

Exclusion Criteria:

* Severe cognitive impairment
* Facial trauma prohibiting headset use
* Physical limitations in facial, neck, upper extremities that hinder use of VR equipment
* Aggression or violence
* Harm to self or others
* Isolation room
* History of seizures or other neurological conditions
* Severe motion sickness
* Active nausea
* Severe visual impairment
* Severe cognitive impairment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-09-14 (Estimated); Study Completion 2026-09-14 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety levels | baseline, immediately after the intervention
  Anxiety levels measured by a Visual Analogue Scale - Anxiety (VAS-A), where participants rate their anxiety in a scale ranging from 0-10, with 0 representing no anxiety to 10 representing extreme anxiety. Higher scores indicate higher anxiety levels.

SECONDARY OUTCOMES:
Change in pain levels | baseline, immediately after the intervention
  Participants will complete the Numerical Rating Pain Scale (NRPS) immediately following each trial, where they rank pain sensitivity on an ordinal scale from 0 = no pain to 10 = worst pain. Higher scores indicate greater or worse pain.
The Perceived Stress Scale | Baseline
  Participants will complete the Perceived Stress Scale-10. It is a five-point Likert-type scale and consists of 10 items. Participants rate each item on a scale ranging from "Never (0)" to "Very often (4)". The total scores range from 0 to 40, and higher scores indicate greater perceived stress.
State-Trait Anxiety Inventory | baseline, immediately after the intervention
  The State-Trait Anxiety Inventory (STAI) is a validated self-report questionnaire consisting of two subscales that measure state anxiety (temporary condition) and trait anxiety (general tendency). Each subscale contains 20 items each, which is rated on a 4-point Likert scale. Scores range from 20 to 80 per subscale, with higher scores indicating greater anxiety, and lower scores indicating no or low anxiety.
Change of Visual Analog Scale for Stress (VAS-Stress) | baseline, immediately after the intervention
  Participants will complete the Visual Analog Scale for Stress (VAS-Stress). Visual analog scale to assess the perceived stress on a horizontal, non-calibrated line of 100 mm, ranging from very low stress (0) to very high stress (100). Higher scores indicate greater stress.
Change in Loneliness as Measured by the UCLA 3-Item Loneliness Scale | baseline, immediately after the intervention
  The UCLA 3-Item Loneliness Scale is a brief, validated self-report questionnaire used to assess subjective feelings of loneliness and social isolation. It consists of three items derived from the original UCLA Loneliness Scale. Each item is rated on a 3-point Likert scale (1 = Hardly Ever, 2 = Some of the Time, 3 = Often), yielding a total score ranging from 3 to 9. Higher scores indicate greater loneliness.
Participant Satisfaction as Measured by a Self-Developed Satisfaction Survey | immediately after the intervention
  Participants will complete the Self-Developed Satisfaction survey. The instrument includes 5 closed-ended items with varying response formats. Two questions are in binary formats, one question is in "Check all that apply" format, one question is on a 5-point Likert scale (1 = Very unlikely, 5=Very Likely) and one is in Numeric rating scales (NRS), response options ranging from 1-2 times to more than 5 times. Responses are coded on a 3-point ordinal scale (1 = 1-2 times, 2 = 3-4 times, 3 = more than 5 times).

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Health Care (SHC), Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No